CLINICAL TRIAL: NCT03307408
Title: Hepatocellular Carcinoma in Patients With a Cirrhosis Due to an Alcoholic or a Non Alcoholic Fatty Liver Disease
Acronym: CHALNA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 16-AOI-12
Record Dates: First submitted 2017-09-15; First posted 2017-10-11 (Actual); Last update posted 2017-10-11 (Actual); Status verified 2017-09

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples, tissu samples, feces samples,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: blood collection — Standard routine practice clinico-biological data will be collected

SUMMARY:
Global prevalence of Non Alcoholic Fatty Liver Diseases (NAFLD) ranges from 22% to 28%.The spectrum of these hepatic abnormalities extends from isolated steatosis to steatohepatitis (Non Alcoholic Steato-Hepatitis, NASH) and steatofibrosis leading to cirrhosis and hepatocellular carcinoma. NAFLD is one of the main causes of cirrhosis and increases the risk of liver-related death and hepatocellular carcinoma (developed in patients with or without cirrhosis). Despite this major public health concern, apart from lifestyle changes, treatment of NAFLD is still elusive as there is lack of efficacious pharmacological treatment. Alcoholic liver diseases are also frequent in Western countries. Alcoholic liver diseases and NAFLD share common pathological lesions and molecular pathways. This is illustrated by the emerging role of abnormalities of the microbiota (dysbiosis) in these 2 diseases leading to the concept of " liver-gut axis ". Whereas the molecular mechanisms responsible for the progression from a "safety" state to NASH or to a severe alcoholic steato-hepatitis are still unclear, hepatic inflammation is a key factor involved in the progression of NAFLD and alcoholic liver disease.

The hypothesis is that cellular and molecular abnormalities and gut dysbiosis could be present in patients with simple steatosis or with steato-hepatitis and could be responsible for the occurrence of hepatocellular carcinoma particularly without cirrhosis.

The main objective is to compare cellular and inflammatory pathways in liver with and without hepatocellular carcinoma in patients with alcoholic or non-alcoholic fatty liver diseases.

ELIGIBILITY:
Group 1

Inclusion Criteria :

* Available social insurance
* Signed consent for the study enrollment
* Age ≥ 18 years

Exclusion Criteria :

* Patients in the group with metabolic fatty liver with hepatocellular carcinoma
* Alcohol consumption ≤ 30 g/d (or 210 g/week) in men and ≤ 20 g/d (or 140 g/week) in women.
* Decision (less than 3 months) to perform a liver biopsy of a tumor suspect of HCC and of adjacent liver in routine practice.
* No systemic HCC treatment in the previous 6 months

Group 2

Inclusion Criteria :

* Available social insurance
* Signed consent for the study enrollment
* Age ≥ 18 years

Exclusion Criteria :

* Patients in the group with metabolic fatty liver without hepatocellular carcinoma
* Alcohol consumption ≤ 30 g/d (or 210 g/week) in men and ≤ 20 g/d (or 140 g/week) in women.
* Decision (less than 3 months) to perform a liver biopsy in routine practice. Liver biopsy will be organized because of one or more liver abnormalities and/or fatty liver seen at liver ultrasound due to the current lack of validated non-invasive marker of inflammation, cellular death and fibrosis in these patients.

Group 3

Inclusion Criteria :

* Available social insurance
* Signed consent for the study enrollment
* Age ≥ 18 years

Exclusion Criteria :

* Patients with an alcoholic liver disease with hepatocellular carcinoma
* Alcohol consumption > 30 g/d (or 210 g/week) in men and > 20 g/d (or 140 g/week) in women.
* Decision (less than 3 months) to perform a liver biopsy of a tumor suspect of HCC and of adjacent liver in routine practice.
* No systemic HCC treatment in the previous 6 months

Group 4

Inclusion Criteria :

* Available social insurance
* Signed consent for the study enrollment
* Age ≥ 18 years

Exclusion Criteria :

* Patients with an alcoholic liver disease without hepatocellular carcinoma
* Alcohol consumption > 30 g/d (or 210 g/week) in men and > 20 g/d (or 140 g/week) in women.
* Decision (less than 3 months) to perform a liver biopsy in routine practice. No systemic HCC treatment in the previous 6 months. Liver biopsy will be organized because of one or more liver abnormalities and/or fatty liver seen at liver ultrasound due to the current lack of validated non-invasive marker of inflammation, cellular death and fibrosis in these patients.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with alcoholic or non-alcoholic fatty liver diseases.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2017-02-28 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Dosage of immunity cells in liver | 8 weeks
  The investigators determine the stage of liver by biochemical, genetic (and immunocytochemistry methods.
Dosage of the inflammatory cells in liver | 8 weeks
  The investigators determine the stage of liver by biochemical, genetic and immunocytochemistry methods.

SECONDARY OUTCOMES:
Dosage of the glucose | 8 weeks
  The investigators determine the genes implicated in oxidative stress, reticulum endoplasmic stress and autophagy .

CONTACTS AND LOCATIONS:
Overall Officials: Rodolphe ANTY, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No